CLINICAL TRIAL: NCT02893046
Title: HCV Care Pathway in Ile-de-France
Acronym: ParcoursVHC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RARS 28
Record Dates: First submitted 2016-08-25; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis C Virus
Keywords: care pathway; hospital- private network; early consultation
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Population at Risk: Population with at least one risk factor of being infected with hepatitis C; MSM population; people in precarious situations and / or attending support from addictions care structures.
  Interventions: Other: No intervention
- Prison population: Proposal of participation to a " consultation arrivants " by the staff of medical units correctional
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The main objective of this research is to evaluate a care pathway adapted to different category populations at risk of being infected with the hepatitis C virus in order to improve both the diagnosis turnaround times and the access to treatment. The aim is to allow a quick and effective access to diagnosis and treatment of HCV by strengthening the city hospital networks, access to early consultations and coordination of medical social actors.

DETAILED DESCRIPTION:
The current estimation of infected persons with chronic hepatitis C in France is over 200 ,000. It appears that prevention, screening, care management, medical and social care of patients can be significantly improved especially among the most vulnerable populations. Indeed, these new HCV infections are mediated by drug-using people, prisoners, migrants, men who have sex with men (MSM) and who are supported too late and without real access to treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and more
* Positive Hepatitis C virus
* Patient having expressed a non-objection to participate in this research

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly screened positive for HCV among private practitioners, screening and diagnostic centers, precarious consultations addictology structures, associations of patients or medical units detention centers.
  Patients already diagnosed positive for HCV but not monitored in a care sector will also be included in the pathway
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients effectively cared divided by number of patients eligible to care. | Year 3

SECONDARY OUTCOMES:
Number of patients cared in the HCV care pathway in Ile-de-France | Year 3
Number of patients effectively treated divided by number of patients eligible to DAA treatment. | Year 3
Delay between HCV diagnosis and early consultation | Year 3

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie DOMINGUEZ, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France